CLINICAL TRIAL: NCT00596063
Title: A Randomized, Single Center, Double Blind, Two Period, Crossover Glucose Clamp Study to Test for Bioequivalence Between Two Recombinant Human Soluble Insulins- Wockhardts Insulin Human Regular for Injection and Novolin R in Healthy Subjects
Brief Title: Comparative Glucose Clamp Study of Wockhardt's Insulin Human Regular for Injection and Novolin R, in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Wosulin R/PK-PD/HV/FDA/07/v1; Not yet created
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus
Keywords: pharmacokinetics; pharmacodynamics; recombinant human insulin; healthy volunteers
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin R (Experimental): Regular insulin for subcutaneous injection (recombinant human insulin), 600nmol, 100 IU
  Interventions: Biological: Wosulin R
- Novolin R (Active Comparator): Regular insulin for injection (recombinant human insulin)
  Interventions: Biological: Novolin R

INTERVENTIONS:
Biological: Wosulin R — Penfill cartridges; Single Dose, 0.2 IU/ kg;
  Arms: Wosulin R
Biological: Novolin R — Penfill cartridges; Single Dose, 0.2 IU/ kg;
  Arms: Novolin R

SUMMARY:
The purpose of this study is the comparative evaluation of the pharmacokinetics and pharmacodynamics of two recombinant regular human insulin injections administered subcutaneously in healthy volunteers under the conditions of euglycemic clamp.

DETAILED DESCRIPTION:
A comparative evaluation of the pharmacokinetics and pharmacodynamics of two recombinant regular human insulin injections administered subcutaneously in healthy volunteers. It is a crossover study. The subjects shall be administered single doses of each insulin during two separate visits under the conditions of euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject.
2. Age ≥ 18 and ≤ 45 years.
3. Body Mass Index (BMI) between 18.0 and 27.0 kg/m2, inclusive.
4. Non-smoker, defined as no nicotine consumption for at least one year.
5. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.).

Exclusion Criteria:

1. Previous participation in this trial or other clinical trials within the last 3 months.
2. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (intrauterine device (IUD) that has been in place for at least 3 months, or sterilization, or the oral contraceptive pill, which should have been taken without difficulty for at least 3 months, an approved hormonal implant).
3. Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with elevated liver enzymes (AST or ALT > 2 times the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit of normal) will not be allowed to enter the trial.
4. Any serious systemic infectious disease during the four weeks prior to the first dose of test drug, as judged by the Investigator.
5. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (haemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
6. History of alcohol or drug abuse.
7. Any positive reaction of drugs of abuse.
8. Hepatitis B or C or HIV positive.
9. Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for oral contraceptives/hormonal implants.
10. Use of any insulin product for therapeutic purposes in the past.
11. Use of non-prescription drugs, except routine vitamins, within 3 weeks prior to the first dose of the test drug. Occasional use of paracetamol is permitted.
12. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
13. Blood donation of more than 500 ml within the last 12 weeks.
14. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
15. Known or suspected allergy to trial product or related products.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to test for bioequivalence based on AUC0-12h and Cmax between Wockhardt's Insulin Human Regular for injection and Novolin® R | Visit 2 & 3

SECONDARY OUTCOMES:
PK endpoints: AUC, tmax and t½ PD endpoints: AUC-GIR, GIRmax and tGIRmax Safety endpoints: AEs, haematology, biochemistry, urinalyses, physical examination, vital signs, ECGs, blood glucose and local tolerability. | Visit 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, M.D, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (2):
- United States (2):
  - Profil Institute for Clinical Research Inc., Chula Vista, California
  - Profil Institute for Clinical Research, Inc., Chula Vista, California